CLINICAL TRIAL: NCT06518369
Title: Analysis of a Preoperative Prehabilitation Program Among Rural Geriatric Patients Compared to Standard of Care
Brief Title: Preoperative Prehabilitation Program For Geriatric Patients in a Rural Healthcare Setting
Status: Completed | Type: Observational
Sponsor: The Guthrie Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 2401-02
Record Dates: First submitted 2024-07-10; First posted 2024-07-24 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Surgery
Keywords: Frailty
MeSH Terms: conditions — Frailty | interventions — Preoperative Exercise

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Non-intervention or standard of care group: 20 Patients who received standard of care
- Prehabilitation Group: 10 patients who take part in a prehabilitation program for 4-6 weeks before surgery
  Interventions: Other: Prehabilitation

INTERVENTIONS:
Other: Prehabilitation — Prehabilitation program for 4-6 weeks before surgery will include:
  * Review of the frailty risk analysis calculator score obtained in the frailty study (#2212-74)
  * Review of lab results including complete blood count, creatinine, albumin, and prealbumin
  * Review of chronic conditions.
  * An office visit or telehealth visit to review instructions on instructions on nutrition, exercise, smoking cessation, and optimization of chronic disease.
  * Drinking surgery immunonutrition drinks twice daily for 5 days before surgery.
  * Educational information and video instruction
  * Weekly phone calls to motivate, ensure adherence, and assess progress.
  * Measurements of hand grip strength and body weight
  Groups: Prehabilitation Group

SUMMARY:
The study will include patients who require elective major abdominal surgery for cancerous or non-cancerous conditions. The goal of the research is to assess the benefit of a prehabilitation program before surgery that includes nutrition, exercise, smoking cessation, and optimization of chronic disease. A group of 10 patients will take part in a prehabilitation program. These patients will be compared to 20 patients who received standard of care.

DETAILED DESCRIPTION:
The study will include patients who require elective major abdominal surgery. The study will compare patients who received standard of care to patients who received a prehabilitation program before surgery.

The prehabilitation program will take place for 4-6 weeks before your surgery and will include:

* Review of frailty risk analysis calculator score obtained in the frailty study (#2212-74)
* Review of lab results including complete blood count, creatinine, albumin, and prealbumin
* Review of chronic conditions
* An office visit or telehealth visit to review instructions on nutrition, exercise, smoking cessation, and optimization of chronic disease.
* Drinking Surgery Immunonutrition shake twice daily for 5 days before surgery.
* Educational information and video instruction
* Weekly phone calls to motivate, ensure adherence, and assess progress.
* Measurements of hand grip strength and body weight

ELIGIBILITY:
Inclusion Criteria:

* Subjects over age 60 who require elective major abdominal surgery

Exclusion Criteria:

* pregnant women

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects over age 60 who require elective major abdominal surgery
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2024-06-18 (Actual); Primary Completion 2024-10-16 (Actual); Study Completion 2025-06-04 (Actual)

PRIMARY OUTCOMES:
Postoperative hospital length of stay | From date of hospitalization until date of hospital discharge, up to 30 days
  Number of days in hospital from date of surgery to date of discharge
Discharge disposition | From date of hospitalization until date of hospital discharge, up to 30 days
  Binary measure of either home or rehabilitation facility

SECONDARY OUTCOMES:
Adverse outcomes after surgery | 30 days after surgery
  Assess adverse outcomes postoperatively
Hospital readmission rates | 30 days after surgery
  Number of times patients are readmitted to the hospital within 30 day of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Georgetson, AGNP-C, Principal Investigator — Robert Packer Hospital Sayre PA
Locations (1):
- Robert Packer Hospital, Sayre, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No